CLINICAL TRIAL: NCT06389552
Title: A Long-term Follow-up Study of FOLFIRINOX Regimen as Adjuvant Therapy in Pancreatic Cancer Patients After Curative Surgery: Multi-center, Prospective
Brief Title: Long-term Observational Study to Evaluate the DFS and OS of Adjuvant FOLFIRINOX Regimen in Pancreatic Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IN_CTP_N01
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Adjuvant Chemotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to evaluate the safety and efficacy of adjuvant FOLFIRINOX regimen in pancreatic cancer patients after curative surgery.

DETAILED DESCRIPTION:
This study is multi-center, prospective, long-term follow-up observational study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 19 at the time of obtaining the informed consent form
* Planning to FOLFIRINOX as adjuvant therapy after pancreatic cancer surgery
* ECOG 0 or 1
* Scheduled to RO or R1 resection
* Organ function capable of chemotherapy

Exclusion Criteria:

* FOLFIRINOX contraindications among the drug approval requirements
* Palliative Therapy
* Experienced toxic reactions or Hypersensitivity reactions of FOLFIRINOX

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 110
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Day 1 to Week 88
  Duration of survival before pancreatic cancer recurrence or death

SECONDARY OUTCOMES:
Overall survival | Day 1 to Week 88
  Duration of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ah Lee, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No